CLINICAL TRIAL: NCT00637013
Title: The Effectiveness and Cost-effectiveness of Operative Versus Non-operative Management of Subacromial Impingement
Brief Title: Operative Versus Non-operative Management of Subacromial Impingement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Academy of Finland (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Juha Paloneva, Md, PhD, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B07103
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial impingement; Shoulder; RCT; Effectiveness; Cost-effectiveness
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acromioplasty (Active Comparator): Acromioplasty + physiotherapy according to a standardized protocol following a 3 months period of active non-operative treatment
  Interventions: Procedure: Acromioplasty
- Physiotherapy (Active Comparator): Physiotherapy according to a standardized protocol following a 3 months period of active non-operative treatment
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Acromioplasty — Arthroscopic or open acromioplasty
  Other Names: Subacromial decompression
  Arms: Acromioplasty
Procedure: Physiotherapy — Physiotherapy according to a standardized protocol
  Other Names: Physical therapy; Non-operative treatment
  Arms: Physiotherapy

SUMMARY:
The study aims at determining the effectiveness and cost-effectiveness of surgical management of subacromial impingement (including partial tears) compared to conservative treatment. The research setting is prospective, randomised, and controlled.

The aim of the study is to search out evidence based data of indications for subacromial decompression. The investigators also aim at offering patients the most efficient and effective treatment and reduce the number of operations that do not have sufficient effectiveness. The data obtained will facilitate developing guidelines for referrals to a specialist when subacromial impingement is suspected.

The investigators hypothesise that there are subgroups of patients suffering from subacromial impingement that benefit from surgery whereas other subgroups are best treated conservatively.

DETAILED DESCRIPTION:
Subgroup analysis:

* age
* sex
* duration of symptoms
* presence of trauma before symptoms
* presence of partial tear
* degenerative findings
* other findings in MRI or arthroscopy
* type of operation
* co-morbidities
* occupation
* pain (VAS)
* objective shoulder function
* activities of daily living

ELIGIBILITY:
Inclusion Criteria:

* age over 35 years old
* duration of symptoms at least three months despite non-operative treatment
* accepts both treatment options (operative and physical therapy)
* must have pain in abduction of the shoulder
* must have painful arc
* must have pain in two of the three isometric tests (0 and 30 degrees of abduction, or external rotation)
* a positive result in the impingement test (a subacromial injection of lidocaine reduces pain)

Exclusion Criteria:

* previous shoulder operations
* too high risk for operation
* any disease or social problem reducing the ability to co-operate
* rheumatoid arthritis
* severe arthrosis of the glenohumeral or acromioclavicular joint
* a full-thickness rotator cuff tear in MRI arthrography
* a progressive malign disease
* adhesive capsulitis
* high-energy trauma before symptoms
* cervical syndrome
* shoulder instability

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain (VAS) and objective shoulder function (Constant score) | 24 months after intervention
  VAS (0 to 100 mm), Constant score (0 to 100 points)

SECONDARY OUTCOMES:
Change in pain (VAS) and objective shoulder function (Constant score) | 3 months after intervention
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 6 months after intervention
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 12 months after intervention
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 5 years after uintervention
  VAS (0 to 100 mm), Constant score (0 to 100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, MD, PhD, Principal Investigator — Central Finland Health Care District, University of Eastern Finland
Locations (3):
- Finland (3):
  - University of Helsinki, Helsinki
  - Central Finland Health District, Jyväskylä
  - Oulu University Hospital, Oulu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brox JI, Gjengedal E, Uppheim G, Bohmer AS, Brevik JI, Ljunggren AE, Staff PH. Arthroscopic surgery versus supervised exercises in patients with rotator cuff disease (stage II impingement syndrome): a prospective, randomized, controlled study in 125 patients with a 2 1/2-year follow-up. J Shoulder Elbow Surg. 1999 Mar-Apr;8(2):102-11. doi: 10.1016/s1058-2746(99)90001-0. PMID 10226960
- [Background] Haahr JP, Ostergaard S, Dalsgaard J, Norup K, Frost P, Lausen S, Holm EA, Andersen JH. Exercises versus arthroscopic decompression in patients with subacromial impingement: a randomised, controlled study in 90 cases with a one year follow up. Ann Rheum Dis. 2005 May;64(5):760-4. doi: 10.1136/ard.2004.021188. PMID 15834056
- [Background] Ketola S, Lehtinen J, Rousi T, Nissinen M, Huhtala H, Konttinen YT, Arnala I. No evidence of long-term benefits of arthroscopicacromioplasty in the treatment of shoulder impingement syndrome: Five-year results of a randomised controlled trial. Bone Joint Res. 2013 Jul 1;2(7):132-9. doi: 10.1302/2046-3758.27.2000163. Print 2013. PMID 23836479
- [Background] Ketola S, Lehtinen J, Arnala I, Nissinen M, Westenius H, Sintonen H, Aronen P, Konttinen YT, Malmivaara A, Rousi T. Does arthroscopic acromioplasty provide any additional value in the treatment of shoulder impingement syndrome?: a two-year randomised controlled trial. J Bone Joint Surg Br. 2009 Oct;91(10):1326-34. doi: 10.1302/0301-620X.91B10.22094. PMID 19794168
- [Background] Haahr JP, Andersen JH. Exercises may be as efficient as subacromial decompression in patients with subacromial stage II impingement: 4-8-years' follow-up in a prospective, randomized study. Scand J Rheumatol. 2006 May-Jun;35(3):224-8. doi: 10.1080/03009740600556167. PMID 16766370
- [Background] Ketola S, Lehtinen J, Elo P, Kortelainen S, Huhtala H, Arnala I. No difference in long-term development of rotator cuff rupture and muscle volumes in impingement patients with or without decompression. Acta Orthop. 2016 Aug;87(4):351-5. doi: 10.1080/17453674.2016.1177780. Epub 2016 Jun 27. PMID 27348693
- [Background] Ketola S, Lehtinen JT, Arnala I. Arthroscopic decompression not recommended in the treatment of rotator cuff tendinopathy: a final review of a randomised controlled trial at a minimum follow-up of ten years. Bone Joint J. 2017 Jun;99-B(6):799-805. doi: 10.1302/0301-620X.99B6.BJJ-2016-0569.R1. PMID 28566400
- [Derived] Cederqvist S, Flinkkila T, Sormaala M, Ylinen J, Kautiainen H, Irmola T, Lehtokangas H, Liukkonen J, Pamilo K, Ridanpaa T, Sirnio K, Leppilahti J, Kiviranta I, Paloneva J. Non-surgical and surgical treatments for rotator cuff disease: a pragmatic randomised clinical trial with 2-year follow-up after initial rehabilitation. Ann Rheum Dis. 2021 Jun;80(6):796-802. doi: 10.1136/annrheumdis-2020-219099. Epub 2020 Dec 3. PMID 33272959
- See also: Clinical Musculoskeletal Diseases Research Group internet pages — http://www.ksshp.fi/musculoskeletalresearch